CLINICAL TRIAL: NCT00159328
Title: Phase 4 Study of Magnetic Resonance Guided Focused Ultrasound Surgery Following Gonadotrophin Releasing Hormone Agonist Treatment for Symptomatic Uterine Fibroids
Brief Title: Efficacy Study of Magnetic Resonance (MR) Guided Focused Ultrasound in the Treatment of Large Fibroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: InSightec-TxSonics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UF008
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Uterine Fibroids
Keywords: Magnetic Resonance Guided Focused Ultrasound; Gonadotrophin Releasing Hormone Agonist; Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

INTERVENTIONS:
Procedure: Magnetic Resonance Guided Focused Ultrasound

SUMMARY:
The purpose of this study is to determine whether ablation of uterine fibroids with MR guided focused ultrasound following 3 months pre-treatment with Gonadotrophin releasing analogues will allow the effective use of this therapy in women with larger fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given consent
* Willing and able to attend all visits
* Minimum age 18 with no desire for future fertility
* Uterine fibroid > 300 cc on MRI
* Normal cervical smear
* Screening symptom score >21
* Pre or peri-menopausal
* Fibroids being device accessible

Exclusion Criteria:

* Pregnancy
* Previous GNRH treatment
* HRT use
* Hormonal Contraception
* Patient on dialysis
* Haematocrit <25
* ASA score > 2
* Severe cerebrovascular disease
* Anticoagulated
* Active pelvic infection or history of PID
* Weight> 250 lbs
* Any contra-indication to MR imaging
* Intolerance to MRI contrast agent
* Unable to remain in prone positions for 3hours
* IUCD
* Abdominal scarring in beam pathway
* Breast feeding
* Non-perfused fibroid on contrast enhanced images

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-03; Study Completion 2006-12

PRIMARY OUTCOMES:
Symptom improvement as judged by validated disease specific questionnaire

SECONDARY OUTCOMES:
Change in fibroid and uterine volume.

CONTACTS AND LOCATIONS:
Overall Officials: wady m gedroyc, Principal Investigator — St Mary's Hospital, Imperial College London.
Locations (1):
- Department of Interventional Magnetic Resonance, St Mary's Hospital, London, United Kingdom

REFERENCES:
- [Background] Hindley J, Gedroyc WM, Regan L, Stewart E, Tempany C, Hynyen K, Mcdannold N, Inbar Y, Itzchak Y, Rabinovici J, Kim HS, Geschwind JF, Hesley G, Gostout B, Ehrenstein T, Hengst S, Sklair-Levy M, Shushan A, Jolesz F. MRI guidance of focused ultrasound therapy of uterine fibroids: early results. AJR Am J Roentgenol. 2004 Dec;183(6):1713-9. doi: 10.2214/ajr.183.6.01831713. PMID 15547216
- [Background] Stewart EA, Gedroyc WM, Tempany CM, Quade BJ, Inbar Y, Ehrenstein T, Shushan A, Hindley JT, Goldin RD, David M, Sklair M, Rabinovici J. Focused ultrasound treatment of uterine fibroid tumors: safety and feasibility of a noninvasive thermoablative technique. Am J Obstet Gynecol. 2003 Jul;189(1):48-54. doi: 10.1067/mob.2003.345. PMID 12861137
- [Background] Tempany CM, Stewart EA, McDannold N, Quade BJ, Jolesz FA, Hynynen K. MR imaging-guided focused ultrasound surgery of uterine leiomyomas: a feasibility study. Radiology. 2003 Mar;226(3):897-905. doi: 10.1148/radiol.2271020395. PMID 12616023